CLINICAL TRIAL: NCT04655651
Title: Effect of Early Identification and Prehabilitation on Postoperative Prognosis in Frail Elderly Undergoing Major Surgeries
Brief Title: Preoperative Frailty and Postoperative Prognosis in the Elderly After Major Surgeries
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.10.26
Record Dates: First submitted 2020-10-26; First posted 2020-12-07 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2022-05

CONDITIONS: Frailty; Age Problem; Surgery
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frailty: patients with a FRAIL Scale of 3 to 5
  Interventions: Other: No intervention
- Non-frailty: patients with a FRAIL Scale of 0 to 2
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention for both groups.

SUMMARY:
Elderly people often have comorbidities. However, there could be a big difference in their health status. Frailty is considered to be relevant to adverse outcomes. Some studies have found that preoperative frailty assessment and comprehensive geriatric assessment (CGA) of the elderly can improve clinical outcomes, but there has been no valid assessment established in China. Therefore it is important to design a research and help to solve this problem.

DETAILED DESCRIPTION:
With an aging population and the improvement of medical technology, the number of elderly patients who need surgery is gradually increasing. Elderly people often have comorbidities, malnutrition, and other conditions leading to an increased risk of anesthesia. What's more, there could be a big difference in the health status of the elderly with the same age. Frailty is considered to be highly prevalent with increasing age and to confer high risk for adverse outcomes. A complete evaluation of elderly patients before surgery may help improve the prognosis. Some studies have found that preoperative frailty assessment and comprehensive geriatric assessment (CGA) of the elderly can improve clinical outcomes, but there has been no valid assessment established in China. In this study, we plan to use a comprehensive preoperative frailty assessment and follow up for 30 days after surgery to explore the effect of preoperative frailty on postoperative complications in the elderly after major surgeries. To better evaluate the postoperative complications, we choose comprehensive complication index (CCI), which integrates all complication of the Clavien-Dindo classification and offers a metric approach to measure morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Aging at least 65 years old.
* Scheduled for major surgery in Peking Union Medical College Hospital .
* Understand and be willing to participate in this research, and can provide written informed consent.

Exclusion Criteria:

* Underwent major surgery within the last month.
* Can't complete the scale evaluation because of lower limb disability or severe knee osteoarthritis and other conditions that affect walking or climbing stairs.
* With mental or neurological disorders and unable to cooperative with investigators.
* Reject to sign the informed consent.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years old who are scheduled for elective major surgery under general anesthesia in Peking Union Medical College Hospital
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
the score of comprehensive complication index(CCI) | 30 days after surgery
  CCI is based on the complication grading by Clavien-Dindo Classification and can be calculated online (https://www.assessurgery.com).

SECONDARY OUTCOMES:
the incidence of postoperative pulmonary complications(PPCs) | 30 days after surgery
  PPCs are a comprehensive evaluation of pulmonary complications. PPCs conclude respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, aspiration pneumonitis, pneumonia, acute respiratory distress syndrome (ARDS), tracheobronchitis, pulmonary oedema, exacerbation of pre-existing lung disease, pulmonary embolus and death.

CONTACTS AND LOCATIONS:
Overall Officials: Li Xu, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
This study will include preoperative evaluations of the elderly scheduled for major surgery. If required, the data could be shared to other researchers.